CLINICAL TRIAL: NCT06305728
Title: Immuno-Positron Emission Tomography, Hyperpolarized C Pyruvate Magnetic Resonance Imaging, and Blood-Based Biomarkers for Early Detection of Pancreatic Adenocarcinoma in Patients With Intraductal Papillary Mucinous Neoplasms
Brief Title: Hyperpolarized C Pyruvate Magnetic Resonance Imaging, and Blood-Based Biomarkers for Early Detection of Pancreatic Adenocarcinoma in Patients With Intraductal Papillary Mucinous Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-367
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cyst
Keywords: Pancreatic Cyst; Memorial Sloan Kettering Cancer Center; 23-367
MeSH Terms: conditions — Pancreatic Cyst | interventions — CA-19-9 Antigen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Risk Pancreatic Cystic Neoplasm: Participants will be diagnosed with a pancreatic cystic neoplasm deemed to be high risk and requiring surgical resection
  Interventions: Diagnostic Test: 89Zr-DFO-HuMab-5B1 immunoPET; Diagnostic Test: HP MRI; Combination Product: Blood assay

INTERVENTIONS:
Diagnostic Test: 89Zr-DFO-HuMab-5B1 immunoPET — Participants who choose to will undergo immunoPET before surgery.
  Other Names: immunoPET
Diagnostic Test: HP MRI — Participants who choose to will undergo HP MRI before surgery.
Combination Product: Blood assay — Will be drawn within 6 weeks of surgery and annually as post operative care
  Other Names: CA19-.9

SUMMARY:
The purpose of this study is for researchers to find ways of detecting pancreatic ductal adenocarcinoma/PDAC early to avoid the invasive procedure of surgery. The study researchers think a combination of imaging and a series of blood tests may be an effective way to detect PDAC early. In this study, researchers will look at whether a combination of the following types of imaging with blood tests can detect PDAC in pancreatic cysts:

* The ImmunoPET scan (immune-positron emission tomography scan) with the imaging agent 89Zr-DFO-HuMab-5B1
* The HP MRI scan (hyperpolarized pyruvate magnetic resonance imaging scan)

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years
* Pancreatic cystic neoplasm deemed to be high risk and requiring surgical resection
* Able to provide informed consent

Exclusion Criteria:

* Pathologic evidence of pancreatic cancer
* Pregnant or breast-feeding patients
* Refusal or inability to tolerate scan (eg anxiety or claustrophobia)
* Inability to lay flat or meet the standard requirements of traditional MRI
* Hepatic function from assays obtained within 6 weeks prior to the study enrollment. For each patient, the upper limit of normal (ULN) value for a particular assay will be defined by the normal reference values of the laboratory that performed the assay

  1. Bilirubin > 1.5 x ULN
  2. AST/ALT > 2.5 x ULN
  3. Albumin < 3 g/dL
  4. GGT > 2.5 x ULN if Alkaline Phosphatase > 2.5 x ULN
* Renal function with Creatinine > 1.5 x ULN or creatinine clearance < 60 mL/min, from assays obtained within 6 weeks prior to study enrollment
* Cardiac: congestive heart failure with New York Heart Association (NYHA) status ≥2, poorly controlled hypertension, a history of clinically significant EKG abnormalities, or myocardial infarction within 6 months of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering (MSK).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2030-03-04 (Estimated); Study Completion 2030-03-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ImmunoPET to identify presence or absence of adenocarcinoma | up to 1 year
  Assess preliminary sensitivity and specificity if the immunoPET is able to identify the presence or absence of adenocarcinoma or high-grade dysplasia in participants who are scheduled to undergo surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Soares, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Weill Cornell Medical Center (Specimen Analysis Only), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org